CLINICAL TRIAL: NCT01709721
Title: A Controlled, Two-Arm, Parallel Group, Randomized Withdrawal Study to Assess the Safety and Efficacy of Hydromorphone Hydrochloride Delivered by Intrathecal Administration Using a Programmable Implantable Pump
Brief Title: Safety and Efficacy Study of Hydromorphone Hydrochloride by Intrathecal Administration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Piramal Critical Care, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CNS-HYD201US
Record Dates: First submitted 2012-08-24; First posted 2012-10-18 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Management of Chronic Pain
Keywords: Hydromorphone; Hydromorphone Hydrochloride; Pain Management; Non-narcotic analgesics
MeSH Terms: conditions — Agnosia | interventions — Hydromorphone; Analgesics, Opioid; Insulin Infusion Systems

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydromorphone Hydrochloride (Randomized/Double-Blind) (Experimental): Subjects on hydromorphone hydrochloride for the duration of therapy.
  Interventions: Drug: Hydromorphone Hydrochloride; Device: Programmable Implantable pump
- Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind) (Active Comparator): Subjects on hydromorphone hydrochloride titrated downward
  Interventions: Drug: Hydromorphone Hydrochloride; Device: Programmable Implantable pump

INTERVENTIONS:
Drug: Hydromorphone Hydrochloride — Opioid for chronic pain
  Other Names: Hydromorphone; Opioid
Device: Programmable Implantable pump — Programmable Implantable pump delivering intrathecal hydromorphone

SUMMARY:
The purpose of this study is to determine the safety and efficacy of hydromorphone hydrochloride by intrathecal administration using a programmable implantable pump.

DETAILED DESCRIPTION:
A Controlled, Two-Arm, Parallel Group, Randomized Withdrawal Study to Assess the Safety and Efficacy of Hydromorphone Hydrochloride Delivered by Intrathecal Administration Using a Programmable Implantable Pump

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included:

1. Subject must be at least 18 years of age and no more than 75 years old.
2. Clinically diagnosed with chronic pain for at least a 6-month period.
3. Subject is presently on intrathecal pain medication and has a SynchroMed II Implantable pump or meets clinical criteria for implantation of a SynchroMed II Implantable pump. Subjects who are naïve to intrathecal therapy, may be enrolled 2-weeks after pump implantation.
4. Subject agrees to sign a Pain Treatment Agreement (Narcotic Contract) limiting narcotic prescriptions to the study physician.
5. Subject must be cognitively intact and, in the opinion of the investigator, capable of participation in the trial.
6. Female subjects of child-bearing potential must agree to use a medically acceptable and effective double-barrier method of birth control.
7. Subjects with existing SynchroMed II Implantable pumps and are reasonably expected to benefit from intrathecal opioid therapy only.
8. Subjects who are capable of receiving an MRI with or without contrast or CT myelogram, if required by the study protocol.
9. Provides written Ethics Committee approved informed consent.
10. Willing to comply with all study procedures and requirements..

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded:

1. Women who are pregnant or are breast-feeding
2. Subjects who have participated in an investigational drug or device trial within 4 weeks prior to enrollment.
3. Subject has any known or suspected allergy to hydromorphone or to the materials of the infusion pump or intrathecal catheter.
4. Subject is scheduled for a pump or catheter replacement within 6 months of their enrollment into the trial.
5. Subject has a history of dependence and abuse of opioids, stimulants, alcohol, or benzodiazepines, as defined by DSM-IV criteria, within the past year (physical dependence on prescribed opioid analgesics is allowed but abuse of opioids according to DSM-IV is not permitted, i.e. opioid addiction for recreational use).
6. Subjects who show signs of active systemic infection.
7. Subjects with a metastatic cancer to the spinal canal or a known central nervous system contraindication to intrathecal therapy.
8. Subject has a condition requiring diathermy procedures.
9. Subject has a life expectancy of less than 12 months.
10. Subject cannot independently comprehend and participate in the required assessments, including responding to the VASPI, Short-form McGill Pain Questionnaire (SF-MPQ), Clinical Opiate Withdrawal Scale (COWS), Subjective Opiate Withdrawal Scale (SOWS), BPI and patient global impression of change (PGIC) measurement tools.
11. Subject is not considered to be medically or psychologically appropriate for pump implantation.
12. Subjects who are unable or unwilling to return to all of the required follow-up visits.
13. Subjects with active implanted devices such as pacemakers, defibrillators, and cochlear implants or other medical device use, if in the opinion of the investigator the device would interfere with the ability to perform an MRI or CT myelogram.
14. As a result of medical review and physical examination, the Investigator considers the subject unfit for the study.
15. Pain located above the shoulders in the head or neck region (e.g. trigeminal neuralgia), central pain syndromes or any other condition in which it is judged to be unlikely that the subject would benefit from intrathecal administration of the drug product.
16. Subjects who have previously been unresponsive to intrathecal hydromorphone therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Rauck, MD, Principal Investigator — The Center for Clinical Research
Locations (1):
- The Center for Clinical Research, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone Hydrochloride (Randomized/Double-Blind): Subjects stay on their current dose of Hydromorphone Hydrochloride administered via intrathecal (IT) pump; depending on the subject's starting dose on hydromorphone hydrochloride, either a 2 mg/mL or 10 mg/mL formulation may be used.
  Hydromorphone Hydrochloride: Opioid for chronic pain
  Device: Programmable Implantable pump delivering intrathecal hydromorphone hydrochloride
- Hydromorphone Titrated Downward/Control (Randomized/Double-Blind): Subjects have their current dose of Hydromorphone Hydrochloride dose titrated downward; administered via Intrathecal pump
  Hydromorphone Hydrochloride: Opioid for chronic pain
  Device: Programmable Implantable pump delivering intrathecal hydromorphone hydrochloride
- Not Randomized (Open Label Only): Enrolled but Not Randomized, dropped out during Open Label phase. Open Label treatment only of their current dose of Hydromorphone Hydrochloride administered via intrathecal (IT) pump; depending on the subject's starting dose on hydromorphone hydrochloride, either a 2 mg/mL or 10 mg/mL formulation may be used.
  Hydromorphone Hydrochloride: Opioid for chronic pain
  Device: Programmable Implantable pump delivering intrathecal hydromorphone hydrochloride
Period: Open Label Phase
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Titrated Downward/Control (Randomized/Double-Blind) | Not Randomized (Open Label Only)
Started (The purpose of the 12-week Open Label Phase of the trial is to titrate subjects to an optimal dose of hydromorphone hydrochloride and demonstrate the ability to maintain adequate pain relief in subjects requiring intrathecal opioid therapy.) | 41 | 40 | 72
Completed | 41 | 40 | 0
Not Completed | 0 | 0 | 72
Not completed — Withdrawal by Subject | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 8
Not completed — Non-compliance With Study Drug | 0 | 0 | 3
Not completed — Investigator Decision | 0 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Changes In The Subject's Condition Render The Subject Unacceptable For Further Treatment | 0 | 0 | 1
Not completed — Inadequate Pain Control | 0 | 0 | 37
Not completed — Other, Specify in text field in database | 0 | 0 | 14
Period: Randomized Phase
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Titrated Downward/Control (Randomized/Double-Blind) | Not Randomized (Open Label Only)
Started (At the end of the Open Label Phase (ie, the 12 week chronic dosing period), subjects who meet criteria for randomization will be assigned to either remain at their current dose of hydromorphone hydrochloride or to have their dose titrated downward (control group) in a blinded fashion.) | 41 | 40 | 0
Completed | 38 | 34 | 0
Not Completed | 3 | 6 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Inadequate Pain Control | 1 | 2 | 0
Not completed — Other, Specify text field in database | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Subjects
Groups:
- Hydromorphone Hydrochloride (Randomized/Double-Blind): Subjects stay on their current dose of Hydromorphone Hydrochloride administered via intrathecal (IT) pump; depending on the subject's starting dose on hydromorphone hydrochloride, either a 2 mg/mL or 10 mg/mL formulation may be used.
  Programmable Implantable pump: Programmable Implantable pump delivering intrathecal hydromorphone
- Hydromorphone Titrated Downward/Control (Randomized/Double-Blind): Subjects have their current dose of Hydromorphone Hydrochloride dose titrated downward; administered via Intrathecal pump
- Total: Total of all reporting groups
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Titrated Downward/Control (Randomized/Double-Blind) | Not Randomized (Open Label Only) | Total
Number analyzed (Participants) | 41 | 40 | 72 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (11.5) | 54.8 (8.3) | 57.1 (9.7) | 55.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 40 | 92
  Male | 14 | 15 | 32 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3 | 6
  Not Hispanic or Latino | 40 | 38 | 69 | 147
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 8
  White | 38 | 36 | 70 | 144
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 72 | 153

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Are Treatment Failures During the Double-blind Randomized Withdrawal Period
Description: Treatment failure during the Randomized Phase is defined as at least one of the following: a) increase of >= 20mm VASPI vs. baseline over 5 days; b) intolerable pain that in investigator's opinion requires intervention; or c) pain-related interventions that violate protocol from Day 84 to Day 119.
  Note: Baseline pain for the randomized phase is defined as the average of the last 5 days with daily pain measurements while on an optimal intrathecal dose of Hydromorphone, between Days 77 and 83 of the open label dosing period.
  Note: A subject who does not have sufficient data for evaluation, drops out for any other reasons that are not listed above or who experiences withdrawal syndrome as identified by COWS > 12 during the randomized phase will not be classified as a treatment failure.
  Note: Analysis period is from beginning of randomization phase (Day 84) to end of study.
Time Frame: 5 weeks [Baseline (Day 84) to Day 119 Visit]
Population: Intent-to-Treat - Randomized Subjects. Subjects in the Open Label Phase of the study who discontinued the study prior to the Randomization Phase and/or did not meet the criteria for randomization are not included in this analysis as they were not randomized to a treatment group.
Measure: Count of Participants; unit: Participants
Groups:
- Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind): Hydromorphone Hydrochloride/Control Titrated Downward
  Hydromorphone Hydrochloride: Opioid for chronic pain
  Programmable Implantable pump: Programmable Implantable pump delivering intrathecal hydromorphone
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
Participants | 18 | 24
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (Randomized/Double-Blind) vs Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind); Superiority of intrathecal hydromorphone hydrochloride as compared to a control arm; Test type: Superiority; p = 0.147, Chi-squared; Pearson's chi-square test

2. Secondary Outcome: Brief Pain Inventory (BPI): Pain Severity, "Worst"
Description: 'Worst' pain experienced in the past 24 hours. Brief Pain Inventory (BPI): Scale: 0 = No Pain, 10 = Pain as bad as you can imagine; a high score indicates a worse outcome.
Time Frame: 5 Weeks [Baseline (Day 84) to Day 119 Visit]
Population: Intent-to-Treat - Randomized. Subjects in the Open Label Phase of the study who discontinued the study prior to the Randomization Phase and/or did not meet the criteria for randomization are not included in this analysis as they were not randomized to a treatment group.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
score on a scale | 5.62 (0.42) | 6.62 (0.43)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (Randomized/Double-Blind) vs Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind); P-value by ANCOVA, with randomization group as the factor and initial parameter value as covariate. Note: For subjects with missing endpoint on Day 119, value is imputed using the Last Observation Carried Forward (LOCF). Note: Baseline for this analysis is the Day 84 visit; Test type: Superiority; p = 0.0342, ANCOVA

3. Secondary Outcome: Brief Pain Inventory (BPI): Pain Severity "Average"
Description: 'Average' pain experienced in the past 24 hours. The Brief Pain Inventory (BPI): Scale: 0 = No Pain, 10 = Pain as bad as you can imagine; a high score indicates a worse outcome.
Time Frame: 5 Weeks [Baseline (Day 84) to Day 119]
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
score on a scale | 4.09 (0.34) | 4.78 (0.35)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (Randomized/Double-Blind) vs Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1642, ANCOVA

4. Secondary Outcome: Brief Pain Inventory (BPI): Pain Severity Summary Measure
Description: Pain severity will be evaluated by rating pain on a scale from 0 (no pain) to 10 (pain as bad as you can imagine) for the 'worst', 'least', and 'average' pain experienced in the past 24 hours, as well as, the pain experienced 'now'. In addition, a calculated mean pain severity score will be based on the sum of all 4 of the pain scores divided by 4. If any of the 4 questions are missing, then the calculated mean pain severity score will be considered missing. High values indicate worse outcome.
Time Frame: 5 Weeks [Baseline (Day 84) to Day 119]
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
score on scale | 4.19 (0.35) | 5.24 (0.36)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (Randomized/Double-Blind) vs Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0160, ANCOVA; ANCOVA, with randomization group as the factor and initial parameter value as covariate

5. Secondary Outcome: Brief Pain Inventory: Interference With Function Summary Measure
Description: Pain interference with daily functioning will be evaluated by rating interference on a scale from 0 (does not interfere) to 10 (completely interferes) for 'general activity', 'mood', 'walking ability', 'normal work', 'relation with other people', 'sleep', and 'enjoyment of life'. A calculated mean pain interference will be based on the sum of non-missing interference questions answered divided by the number of questions answered. The mean should be set to missing if fewer than 4 pain interference questions are answered. A high score is worse.
Time Frame: 5 Weeks [Baseline (Day 84) to Day 119]
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
score on scale | 3.76 (0.44) | 5.54 (0.45)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (Randomized/Double-Blind) vs Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0007, ANCOVA; ANCOVA, with randomization group as the factor and initial parameter value as covariate

6. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ): Summary Score
Description: The SF-MPQ consists of a 15 item pain rating index. The severity of each item will be scored as None (0), Mild (1), Moderate (2), or Severe (3). The total SF-MPQ score is the sum of the severity scores for each item. The total score can range from 0 to 45; high score is worse.
Time Frame: 5 Weeks [Baseline (Day 84) to Day 119]
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale, summed across 15 quest
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
score on a scale, summed across 15 quest | 11.05 (1.53) | 16.95 (1.55)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (Randomized/Double-Blind) vs Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0088, ANCOVA — ANCOVA, with randomization group as the factor and initial parameter value as covariate

7. Secondary Outcome: Time to Rescue Medication After Randomization (Days)
Description: The number of days to rescue will be calculated by calculating the number of hours between the time of randomization and the time of rescue. The number of hours will then be divided by 24 to obtain the number of days.
Time Frame: 5 Weeks [Baseline (Day 84) to Day 119]
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
days | 28.85 (6.32) | 24.35 (9.67)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (Randomized/Double-Blind) vs Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind); Test type: Superiority; p = 0.011, Log Rank — Log-rank test for Kaplan-Meier Estimate of Time to Rescue (days)

8. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC rating represents observed changes (if any) from the subject's Baseline Visit in activity limitations, symptoms, emotions, and overall quality of life, related to the subject's painful condition. Change is rated on a 7-point Likert-type scale from 1 (no change) through 7 (a great deal better). High score is better outcome.
Time Frame: 5 Weeks [Baseline (Day 84) to Day 119 / Treatment Failure]
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
score on a scale | 4.95 (1.70) | 3.73 (2.04)
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (Randomized/Double-Blind) vs Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind); P-value by the Cochran-Mantel-Haenszel mean score test (using equally spaced scores); Test type: Superiority; p = 0.0335, Cochran-Mantel-Haenszel

9. Secondary Outcome: Oral Opioid Supplement Consumption
Description: Total consumption (mg) = The total number of milligrams consumed of any oral opioid product from Day 84 (Baseline) through the end of study will be calculated for each subject.
Time Frame: 5 Weeks [Baseline (Day 84) to Day 119]
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
milligrams (mg) | 6916.88 (14102.91) | 1732.84 (5984.53)

10. Secondary Outcome: Time to Rescue - Rescue Medication Given
Description: Number of subjects with rescue medication given
Time Frame: 5 Weeks [Baseline (Day 84) to Day 119]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind)
Number analyzed (Participants) | 41 | 40
Participants | 16 | 27
Statistical Analysis 1: Comparison: Hydromorphone Hydrochloride (Randomized/Double-Blind) vs Hydromorphone Hydrochloride Titrated Downward/Control (Randomized/Double-Blind); Test type: Superiority — Pearson's chi-square test; p = 0.010, Chi-squared — Pearson's chi-square test

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Includes all subjects who have study medication loaded into their intrathecal pump (ie, any exposure to hydromorphone hydrochloride).
Groups:
- Not Randomized (Open Label Only): Enrolled but not randomized [Entered Open Label Phase includes visits from Day 1 until date of randomization (Day 84)]
- All Subjects: Total serious adverse events from Day 1 through end of study
Arm/Group | Hydromorphone Hydrochloride (Randomized/Double-Blind) | Hydromorphone Titrated Downward/Control (Randomized/Double-Blind) | Not Randomized (Open Label Only) | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40 | 0/72 | 0/153
Serious Adverse Events (participants affected / at risk) | 2/41 | 6/40 | 9/72 | 17/153
Other Adverse Events (participants affected / at risk) | 35/41 | 36/40 | 56/72 | 127/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone Hydrochloride (Randomized/Double-Blind) (N=41) | Hydromorphone Titrated Downward/Control (Randomized/Double-Blind) (N=40) | Not Randomized (Open Label Only) (N=72) | All Subjects (N=153)
Akathisia (Nervous system disorders) | 0 | 1 | 0 | 1
Basal Ganglia Stroke (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Drug Withdrawal Syndrome (General disorders) | 0 | 2 | 0 | 2
Drug Intolerance (General disorders) | 0 | 0 | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 1 | 1
Implant Site Abscess (Infections and infestations) | 0 | 0 | 1 | 1
Implant Site Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Incision Site Infection (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1 | 2
Angina Unstable (Cardiac disorders) | 0 | 1 | 0 | 1
Oesophageal Achalasia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hydromorphone Hydrochloride (Randomized/Double-Blind) (N=41) | Hydromorphone Titrated Downward/Control (Randomized/Double-Blind) (N=40) | Not Randomized (Open Label Only) (N=72) | All Subjects (N=153)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 9 | 7 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 6 | 11
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 5 | 5 | 10
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 8
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 4
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Drug Withdrawal Syndrome (General disorders) | 3 | 11 | 8 | 22
Pain (General disorders) | 3 | 5 | 3 | 11
Oedema Peripheral (General disorders) | 3 | 1 | 3 | 7
Chills (General disorders) | 1 | 2 | 1 | 4
Oedema (General disorders) | 2 | 2 | 0 | 4
Chest Pain (General disorders) | 0 | 2 | 1 | 3
Asthenia (General disorders) | 0 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 12 | 15 | 8 | 35
Diarrhoea (Gastrointestinal disorders) | 4 | 10 | 3 | 17
Vomiting (Gastrointestinal disorders) | 3 | 7 | 2 | 12
Constipation (Gastrointestinal disorders) | 2 | 5 | 1 | 8
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Headache (Nervous system disorders) | 4 | 4 | 6 | 14
Somnolence (Nervous system disorders) | 2 | 1 | 4 | 7
Sciatica (Nervous system disorders) | 0 | 2 | 3 | 5
Lethargy (Nervous system disorders) | 1 | 2 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 2
Bronchitis (Infections and infestations) | 3 | 2 | 3 | 8
Gastroenteritis Viral (Infections and infestations) | 1 | 3 | 2 | 6
Sinusitis (Infections and infestations) | 3 | 1 | 2 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 1 | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 8
Anxiety (Psychiatric disorders) | 1 | 4 | 2 | 7
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 6
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 4
Joint Injury (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 3
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 3 | 0 | 4
Hypertension (Vascular disorders) | 1 | 3 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT01709721/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT01709721/SAP_001.pdf